CLINICAL TRIAL: NCT05162170
Title: Primary Mediastinal Large B-cell Lymphoma (PMBCL): Multicenter Retrospective Study by the Fondazione Italiana Linfomi.
Brief Title: Primary Mediastinal Large B-cell Lymphoma (PMBCL): Multicenter Retrospective Study
Status: Completed | Type: Observational
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Other Study IDs: FIL_PMBCL
Record Dates: First submitted 2021-11-26; First posted 2021-12-17 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Primary Mediastinal Large B-cell Lymphoma (PMBCL)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Primary Mediastinal large B-Cell Lymphoma (PMBCL): The present study consists of a retrospective multicenter collection of series of consecutive patients diagnosed with PMBCL over the relevant time period (13 years, from 2007 to 2019 included).

SUMMARY:
The present study consists of a retrospective multicentric collection of all consecutive patients with PMBCL diagnosed over the time period considered (13 years, from 2007 to 2019 inclusive).

DETAILED DESCRIPTION:
The study was initially set up as a spontaneous, non-profit study, with ARNAS Garibaldi of Catania (PI Dr Ugo Consoli) as the proposer. Subsequently, the project was expanded to include additional centres belonging to the Italian Lymphoma Foundation, which became the promoter in collaboration with ARNAS Garibaldi of Catania. The information collected is aimed at verifying the application in a "real world" context of the PMBCL diagnosis and therapy protocols suggested in the guidelines and at checking whether they produce results in line with those expected.

The therapies considered for the I line of treatment are those described in the literature for the pathology under consideration:

* R-CHOP14; R-CHOP21 and R-CHOP like, (R-CHOP: rituximab - cyclophosphamide, doxorubicin, vincristine, prednisone)
* R-VACOPB, R-MACOPB and R-VACOPB like, MACOPB like, (R-VACOP-B: Rituximab - etoposide, doxorubicin, cyclophosphamide, vincristine, prednisone, bleomycin. R-MACOP-B: Rituximab - methotrexate, doxorubicin, cyclophosphamide, vincristine, prednisone, bleomycin)
* R-DA-EPOCH ed R-EPOCH like (DA-R- EPOCH: Dose Adjusted - Rituximab - Etoposide, Prednisone, Vincristine, Cyclophosphamide, Doxorubicin)

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients treated in the centre during the period considered
* Age>=18 years
* Histological diagnosis of PMBCL
* Signature of "Informed Consent" to participate in the study (if applicable)
* Treatment according to local practice
* Diagnosis between 01 January 2007 and 31 December 2019

Exclusion Criteria:

- The exclusion criteria, being an observational study, are focused and limited to excluding cases with a non-compliant histological diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients newly diagnosed with PMBCL between 01 January 2007 and 31 December 2019 attending participating centres.
Sampling Method: Non-Probability Sample
Enrollment: 633 (Actual)
Dates: Start 2019-10-02 (Actual); Primary Completion 2022-12-05 (Actual); Study Completion 2025-07-11 (Actual)

PRIMARY OUTCOMES:
Rate of primary/early refractory disease | The endpoint will be evaluated from the beginning to the end of the study (up to 24 months)
  The study aims to evaluate the rate of primary/early refractory disease (Primary mediastinal large B-cell lymphoma)
Overall response rate (ORR) | The endpoint will be evaluated from the beginning to the end of the study (up to 24 months)
  Overall Response Rate is defined as the percentage of patients in complete remission or in partial remission
Complete response rate (CRR) | The endpoint will be evaluated from the beginning to the end of the study (up to 24 months)
  The Complete Response Rate is defined as the percentage of patient in Complete Remission
Frequency of administration of mediastinal radiation therapy | four months after completion of chemotherapy
  Analyze the frequency of administration of mediastinal radiation therapy in patients affected by primary mediastinal large B-cell lymphoma
Progression Free Survival (PFS) | The endpoint will be evaluated from the beginning to the end of the study (up to 24 months)
  The length of time during and after the treatment that patients live with the disease, but it does not get worse. Progression-Free Survival (PFS) will be defined from the date of starting therapy and the date of disease progression, relapse or death from any cause.
Overall Survival (OS) | The endpoint will be evaluated from the beginning to the end of the study (up to 24 months)
  Overall Survival, the percentage of patients alive, is defined from the start date of therapy to the date of death from any cause.

SECONDARY OUTCOMES:
Acute toxicity | The endpoint will be evaluated from the beginning to the end of the study (up to 24 months)
  Analyze incidence and type of acute toxicity (haematological and extra haematological toxicity)
Long-term toxicity | The endpoint will be evaluated from the beginning to the end of the study (up to 24 months)
  Analyze incidence and type of long-term toxicity (cardiological toxicity and second tumors)

CONTACTS AND LOCATIONS:
Overall Officials: Ugo Consoli, Principal Investigator — U.O.C Ematologia, ARNAS Garibaldi; P.O. Garibaldi - Nesima, Catania.
Locations (40):
- Italy (40):
  - U.F. Oncoematologia, IOM (Istituto Oncologico del Mediterraneo), Viagrande, Catania
  - SC Ematologia, A.O. SS. Antonio e Biagio e Cesare Arrigo, Alessandria
  - Clinica di Ematologia, AOU Ospedali Riuniti, Ancona
  - Azienda Ospedaliera S.Giuseppe Moscati - S.C. Ematologia e Trapianto emopoietico, Avellino
  - Divisione di Oncologia e dei Tumori immuno-correlati, IRCCS Centro di Riferimento Oncologico di Aviano, Aviano
  - U.O. Ematologia con Trapianto, AOU Policlinico Consorziale, Bari
  - U.O.C. Ematologia - IRCCS Istituto Tumori Giovanni Paolo II, Bari
  - Ematologia, Ospedale "Monsignor Raffaele Dimiccoli", Barletta
  - Istituto di Ematologia "Seragnoli", Policlinico S.Orsola-Malpighi, Bologna
  - Ematologia, ASST Spedali Civili di Brescia, Brescia
  - U.O. Ematologia e Trapianti di Midollo, Ospedale Antonio Perrino, Brindisi
  - SC Ematologia e CTMO, Ospedale Businco, Cagliari
  - Arnas Nuovo Ospedale Garibaldi Nesima, Catania
  - Ematologia, Azienda Ospedaliero - Universitaria Policlinico - Vittorio Emanuele Presidio Ospedale Ferrarotto, Catania
  - UOC Ematologia, Azienda Ospedaliera di Cosenza, Cosenza
  - Unitа funzionale di Ematologia, Azienda Ospedaliera Universitaria Careggi, Florence
  - Ematologia, Ospedale Vito Fazzi, Lecce
  - Ematologia, Ospedale Madonna delle Grazie, Matera
  - SC Ematologia, Azienda Ospedali Riuniti Papardo-Piemonte, Messina
  - Ematologia, Fondazione IRCCS Istituto Nazionale dei Tumori di Milano, Milan
  - Divisione Ematoncologia, IEO Istitito Europeo di Oncologia, Milan
  - SC Ematologia, ASST Grande Ospedale Metropolitano Niguarda, Milan
  - UOC Ematologia Oncologica, Istituto Nazionale Tumori - IRCCS Fondazione G. Pascale, Napoli
  - Istituto Oncologico Veneto I.R.C.C.S., Padua
  - Ematologia, AOU Policlinico Giaccone, Palermo
  - Divisione di Ematologia, A.O. Ospedali Riuniti Villa Sofia-Cervello, Palermo
  - Oncoematologia e TMO Dip. Oncologia, Casa di Cura La Maddalena, Palermo
  - Azienda Ospedaliera Universitaria Pisana - U.O. Ematologia, Pisa
  - Ematologia, Grande Ospedale Metropolitano Bianchi Melacrino Morelli, Reggio Calabria
  - Ematologia, Azienda Unitа Sanitaria Locale-IRCCS - Arcispedale Santa Maria Nuova, Reggio Emilia
  - Ematologia, Ospedale S. Camillo, Roma
  - Istituto Ematologia -Dipartimento di Medicina Traslazionale e di Precisione,Policlinico Umberto I - Universitа "La Sapienza", Roma
  - Ematologia, Universitа Cattolica S. Cuore, Roma
  - UO Ematologia, Istituto Clinico Humanitas, Rozzano
  - UO Ematologia, Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - SC Ematologia, Ospedale "S.G. Moscati", Taranto
  - Azienda Ospedaliera Santa Maria - S.C. Oncoematologia, Terni
  - Ematologia Universitaria, A.O.U. Citta della Salute e della Scienza di Torino, Torino
  - SC Ematologia, A.O.U. Citta della Salute e della Scienza di Torino, Torino
  - UO Ematologia, AOU Integrata di Verona, Verona